CLINICAL TRIAL: NCT06562621
Title: Clinical Study on the Safety and Efficacy of Novel Oncolytic Virus in the Treatment of Recurrent Malignant Glioma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Beijing Neurosurgical Institute (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CFH2020-1-1071
Record Dates: First submitted 2024-08-13; First posted 2024-08-20 (Actual); Last update posted 2024-08-20 (Actual); Status verified 2024-08

CONDITIONS: Glioblastoma Multiforme; Gliomas, Malignant
MeSH Terms: conditions — Glioblastoma; Glioma | interventions — Oncolytic Virotherapy; Flucytosine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- ON-01/ONF (Experimental): ON-01: 1ml intratumoral injection of ON-01. ONF: 100 mg/kg/day orally after operation for 20 consecutive days.
  Interventions: Biological: ON-01; Drug: ONF

INTERVENTIONS:
Biological: ON-01 — ON-01 consists of a yeast cytosine deaminase (CD) gene. The CD gene converts the antifungal 5-flurocytosine (5-FC) to the anticancer drug 5-FU in cells that have been infected by ON-01.
  Other Names: Oncolytic virus; Herpes simplex virus
Drug: ONF — ONF is an extended-release formulation of flucytosine.
  Other Names: Flucytosine; 5-FC; 5-Fluorocytosine

SUMMARY:
Glioma is the most common intracranial tumor. Among them, malignant glioma shows diffuse and infiltrating growth. Although it is given a comprehensive treatment such as surgery, radiotherapy and chemotherapy, it is prone to relapse, and there is an urgent need to explore new treatment methods. Oncolytic virus is currently the world's most cutting-edge treatment of glioma. On the basis of previous research on glioma and oncolytic virus (HSV-1), an engineered new oncolytic virus ON-01 containing CD gene has been constructed. In vitro and in vivo animal experiments have found that it has a good therapeutic effect on malignant glioma, and it has been approved by the ethics committee of Tiantan Hospital for its clinical research. This project intends to study the safety and effectiveness of ON-01 in the clinic on the basis of pre-clinical trials and preclinical research, clarify the oncolytic mechanism of ON-01 in the treatment of malignant glioma, and explore the dissolution of brain glioma. The new strategy of tumor virus treatment lays a theoretical foundation for the clinical promotion and application of ON-01 and product transformation.

ELIGIBILITY:
Inclusion Criteria:

1. Patients has given written informed consent；
2. Age is between 18 years old and 75 years old, inclusive;
3. Patients must have histologically or cytologically confirmed Glioblastoma, anaplastic astrocytoma, anaplastic oligodendroglioma, anaplastic oligodendrocyte-glioma;
4. Residual lesion must be ≥1.0 cm in diameter as determined by MRI;
5. Karnofsky Performance Status ≥70%;
6. Patients must have normal organ and marrow function. Absolute neutrophil count: ≥ 1,500/mm3, Hemoglobin>10 g/dL platelets: >100,000/mm3, total bilirubin< 1.5 ×ULN; AST(SGOT)(aspartate aminotransferase)/ALT(SGPT)(alanine aminotransferase): <2.5 X institutional upper limit of normal; Serum creatinine < 1.5 ×ULN, and normal heart function;
7. Good compliance: can actively cooperate with doctors' treatment and follow-up survey;
8. Females of childbearing potential must not be pregnant; this will be confirmed by a negative serum pregnancy test within 7 days prior to starting study treatment and must use a birth control method in addition to barrier methods (condoms).

Exclusion Criteria:

1. Pregnant or lactating women;
2. Prior history of encephalitis, multiple sclerosis, or other CNS infection;
3. Herpes simplex virus infection active period;
4. Patients with a history of organ transplantation or waiting for an organ transplant;
5. Uncontrollable infectious diseases or other serious diseases such as HIV positive;
6. Severe pulmonary, cardiac or other systemic disease, specifically: Including active infections, uncontrolled high blood pressure, unstable angina pectoris, angina pectoris that began to develop within the last 3 months, congestive heart failure, myocardial infarction that occurred within the first 12 months of enrollment, requiring serious;medical treatment Arrhythmia, liver, kidney failure, etc.;
7. Patients with systemic autoimmune disease or immunodeficiency disease;
8. Patients with severe allergies;
9. Patients with chronic diseases requiring long-term immunologic preparation or glucocorticoid therapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-08-01 (Actual); Primary Completion 2022-08-01 (Actual); Study Completion 2024-03-01 (Actual)

PRIMARY OUTCOMES:
Long term safety follow up | From study entry up to 5 years
  The short-term adverse reactions of the subjects during hospitalization after receiving stereotactic injection of the oncolytic virus ON-01 will be recorded, and the incidence of these adverse reactions will be statistically analyzed. The short-term adverse reactions include: nausea, altered mental status, fever, pyramidal tract syndrome, flush face, epilepsy, anemia, leukopenia, thrombocytopenia, hyponatremia, hypokalemia, hypocalcemia, arrhythmia. These adverse reactions will be classified into four grades according to their severity. Within two weeks, a specialized neurosurgeon will conduct a clinical examination on the subjects to assess their motor, sensory, and language functions. Detailed post-injection treatment of each patient was recorded. Patients unwilling to accept or failed to complete the treatment due to safety or economic reasons were stratified as incomplete treatment group.

SECONDARY OUTCOMES:
Overall survival in days from the initial ON-01 administration on parent study to the date of death. | From initial ON-01 administration to death of last patient alive for up to 5 years.
  Overall survival (OS) defined as the duration from the date of stereotactic biopsy to the date of death or last follow up. At baseline, all patients underwent a thorough examination including blood cell counts, blood chemical analysis (including hepatic and renal function). Tumor sample of each patient was examined by 3 independent neuro-pathologists. Patients with the diagnosis other than recurrent GBM in paraffin section were excluded from the study. On the tenth day after injection, an enhanced MRI was carried out to evaluate tumor response. Tumor and residual tumor size was approximately estimated using the sum of the products of the largest perpendicular diameters of enhanced lesion. The clinical, operative, and hospitalization records were retrospectively reviewed. The Karnofsky Performance scale (KPS) score was used to describe patients' functional status.
Progression-free survival in days from the initial ON-01 administration on parent study to confirmed disease progression or death from any cause. | from initial ON-01 administration to time of progression or death of any cause for up to 5 years.
  Progression-free survival (PFS) refers to the length of time after a patient receives treatment with the oncolytic virus ON-01 during which the size of the glioma tumor either decreases or does not increase further on imaging. It is used as an indicator to assess the effectiveness of the oncolytic virus treatment. A longitudinal follow-up was planned for each patient at the following time points: the tenth day after injection, monthly thereafter, or whenever symptoms suggesting tumor relapse occurred. Each follow-up included an enhanced MRI to detect possible asymptomatic tumor recurrence and a blood test to find adverse events. Undetermined MRI scan were carefully reviewed by a senior neurosurgeon and neuroradiologist to differentiate tumor recurrence and radiation induced encephalic necrosis. If necessary, serial of MRI scans or positron emission tomography (PET) were performed.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Tiantan Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No